CLINICAL TRIAL: NCT00108589
Title: S-Adenosylmethionine Therapy for Non-Alcoholic Steatohepatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CLIN-014-03S
Record Dates: First submitted 2005-04-15; First posted 2005-04-18 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2007-05

CONDITIONS: Hepatitis
Keywords: s-adenosylmethionine; fatty liver; obesity; Non-alcoholic steatohepatitis
MeSH Terms: conditions — Hepatitis; Fatty Liver; Obesity; Non-alcoholic Fatty Liver Disease | interventions — S-Adenosylmethionine

INTERVENTIONS:
Drug: S-adenosylmethionine

SUMMARY:
The purpose of this study is to examine the effect of S-adenosylmethionine therapy in those patients with non-alcoholic liver disease in the form of steatohepatitis (NASH). This will be accomplished by development of a database of these patients, all of whom will have biopsy documented NASH. A placebo controlled trial will then examine the effect of S-adenosylmethionine over time on clinical outcome in these patients. It is expected that this agent will slow or halt the progression of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Men with biopsy proven non-alcoholic steatohepatitis from the liver disease clinic or referred from other physicians from the VAMC-Louisville.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-01; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Locations (1):
- VA Medical Center, Louisville, Kentucky, United States